CLINICAL TRIAL: NCT07402577
Title: Brief Title Mechanisms of Cancer-Related Pain and Opioid Use Among Adolescents and Young Adult Sarcoma Survivors: Pilot Feasibility Study
Status: Not yet recruiting | Type: Observational
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: University at Buffalo (Other)
Responsible Party: Sponsor
Other Study IDs: I-4720925
Record Dates: First submitted 2026-01-28; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Sarcoma; Childhood Sarcoma of Soft Tissue
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non Intervention Study — Non intervention study

SUMMARY:
This study generates information on the feasibility and acceptability of a 3-month ecological momentary assessment (EMA) protocol to assess chronic pain and opioid use in adolescent and young adult (AYA) sarcoma survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the feasibility and acceptability of a 3-month EMA protocol in AYA sarcoma survivors.

II. Quantify variability in pain and opioid use over a 3-month period for AYA sarcoma survivors.

III. Identify associations between biopsychosocial mechanisms (e.g., pain beliefs, worry) and pain and opioid use outcomes.

OUTLINE: This is an observational study.

Patients complete baseline questionnaires, daily EMA surveys and an interview on study.

ELIGIBILITY:
Inclusion Criteria:

* All genders between the ages of 12-24 (inclusive) at sarcoma diagnosis.
* Any age < 70 at the time of study enrollment.
* No evidence of disease and/or enrolled in survivorship care.
* Clinically meaningful pain related to disease or its treatments at baseline (defined as 3 or greater on a 0-10 Numerical Rating Scale).
* Willing to attend the baseline appointment in person.
* Access to internet-capable smartphone.
* Access to internet on an occasional basis.
* Willing and able to complete Ecological Momentary Assessments (EMAs) on internet-capable smartphone for a 3-month period after enrollment.
* Ability to understand and provide informed consent/assent.

Exclusion Criteria:

* * Currently receiving active cancer-directed therapy.

  * Unable to read or fluently speak English.
  * Determined by clinical staff to have preexisting or cancer-associated cognitive impairment that could interfere with study participation.
  * Acutely suicidal (e.g. intent or plan) or, with unstable medical or psychiatric condition verified by licensed study staff.
  * Characteristics related to inability to complete the study protocol.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients younger than 70 years old who were diagnosed with sarcoma between the ages of 12-24 and have no evidence of disease and/or are enrolled in survivorship care.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-02-22 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment | Up to 12 months
  Feasibility of recruitment will be based on number eligible per medical record
Feasibility of assessment | Up to 12 months
  will be indexed by number completing 80% of EMA assessments
Feasibility of recruitment | up to 12 months
  will be indexed by number attending baseline interview
Feasibility of recruitment | Up to 12 months
  will be indexed by retention throughout EMA period
Reasons for nonparticipation | UP to 12 months
  Semi structured qualitive interviews will focus on factors that influenced participation
Acceptability of EMA Study Design | Up to 12 months
  self-reported difficulty of participating in daily EMA surveys (0-19) .
Acceptability of EMA Design | Up to 12 months
  Acceptability of the protocol will be assessed by responses on the System Usability Scale - A 10 question scale from 1 to 5 with 1 being strongly disagree and 5 being strongly agree.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Rogers, Principal Investigator — Roswell Park

IPD SHARING:
Plan to Share IPD: Undecided